CLINICAL TRIAL: NCT06553339
Title: A Phase I Study of HS-10516 in Patients With VHL Syndrome Associated Tumors，to Investigate Safety, Tolerance, Pharmacokinetic and Efficacy
Brief Title: A Study of HS-10516 in Patients With VHL Syndrome Associated Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HS-10516-102
Record Dates: First submitted 2024-08-12; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Von Hippel Lindau-Deficient Clear Cell Renal Cell Carcinoma
Keywords: Von Hippel Lindau Syndrome; VHL Syndrome; RCC; pNET; CNS hemangioblastoma
MeSH Terms: conditions — von Hippel-Lindau Disease; Neuroectodermal Tumors, Primitive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phase Ia dose escalation arm (Experimental): Participants will be assigned to pre-specified dose level to identify the MTD/MAD of HS-10516.
  Interventions: Drug: Oral HS-10516
- Phase Ib dose expansion arm 1 (Experimental): Participants with VHL Syndrome associated RCC, whose lesions diameter ≤ 3 cm.
  Interventions: Drug: Oral HS-10516
- Phase Ib dose expansion arm 2 (Experimental): Participants with VHL Syndrome associated RCC, who could not be included in arm 1.
  Interventions: Drug: Oral HS-10516
- Phase Ib dose expansion arm 3 (Experimental): Participants with VHL Syndrome associated non-RCC tumors.
  Interventions: Drug: Oral HS-10516

INTERVENTIONS:
Drug: Oral HS-10516 — Oral HIF-2α inhibitor

SUMMARY:
The aim of the Phase Ia portion is to identify the maximum tolerated dose or maximum acceptable dose MTD/MAD of HS-10516. The phase Ib portion will evaluate the preliminary efficacy of HS-10516 in patients with VHL Syndrome Associated Tumors.

DETAILED DESCRIPTION:
This is a Phase Ia/Ib open label multicenter study of HS-10516 in Chinese patients aged 18 years or older with VHL Syndrome Associated Tumors. HS-10516 as a single agent, is administrated orally once daily. The aim of phase Ia, a dose escalation study, is to identify the MTD/MAD of HS-10516. The goal of Phase Ib, a dose expansion study, is to evaluate the safety, pharmacokinetics and antitumor efficacy of HS-10516.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female from 18 to 80 year-old
2. Patients with advanced clear cellrenal cell carcinoma or von Hippel-Lindau Syndrome associated tumors
3. Has an Eastern Cooperative Oncology Group performance status of 0-1
4. Has a life expectancy of ≥ 12 weeks
5. Should use adequate contraceptive measures throughout the study
6. Females subject must not be pregnant at screening
7. Has the ability to understand and willingness to sign a written informed consent before the performance of the study.

Exclusion Criteria:

1. Recieved or being received treatment as follows:

   1. Hypoxia-induced factor inhibitors
   2. Traditional Chinese medicine indicated for tumors within 2 weeks prior to the first dose of study treatment.
   3. Cytotoxic chemotherapeutic drugs, investigational drugs or other systematic anti-tumor therapies within 3 weeks before the first dose of study treatment
   4. Colony-stimulating factors (CSFs) within 4 weeks before the first dose of study treatment
   5. Local radiotherapy within 2 weeks prior to the first dose of study treatment; more than 30% of bone marrow radiotherapy or large-area irradiation within 4 weeks before the first dose of study treatment.
   6. Major surgery within 4 weeks prior to the first dose of study treatment.
2. Has a pulse oximetry reading less than 92% at screening, requires intermittent supplemental oxygen, or requires chronic supplemental oxygen
3. Has failed to recover from a ≥ grade 2 adverse event due to prior anti-tumor therapy
4. Has another malignancy or a history of another non-VHL syndrome associated malignancy
5. Has inadequate bone marrow reserve or organ dysfunction
6. Has a clinically significant bleeding events or tendency within 1 month prior to the first dose of study treatment
7. Has severe infections within 4 weeks prior to the first dose of study treatment
8. Has digestive system diseases may influencing ADME of study drug
9. Has a history of severe hypersensitivity reaction, or proven allergic to HS-10516 or its metabolin
10. Has any disease or condition would compromise subject safety or interfere with study assessments by investigator's decision

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Phase Ia: MTD/MAD of HS-10516 | Approximately 2 months
  Maximum Tolerated Dose or Maximum Acceptable Dose determined by the Number of Participants with Dose Limiting Toxicity (DLT) events during the DLT monitoring period (first 35 days of dosing) in the Dose Escalation Phase
Phase Ib: Objective Response Rate (ORR) by Independent Review Committee (IRC) | Approximately 1 year
  ORR defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. ORR will be assessed by IRC.

SECONDARY OUTCOMES:
The Number of Participants with Adverse Events | Approximately 2 years
  An adverse event (AE) is defined as any untoward medical occurrence in a patient and which does not necessarily have a causal relationship with this treatment. The investigator assessed the relationship of each event to the use of study drug as either probably related, possibly related, probably not related or not related.
Observed maximum plasma concentration (Cmax) of HS-10516 | Approximately 2 months
  Cmax will be obtained following administration of the first dose of HS-10516 during first 2 cycles.
Time to reach maximum plasma concentration (Tmax) of HS-10516 | Approximately 2 months
  Tmax will be obtained following administration of the first dose of HS-10516 during first 2 cycles.
Area under plasma concentration versus time curve from zero to last sampling time (AUC0-t) following the first dose of HS-10516 | Approximately 1 year
  Area under the plasma concentration versus time curve from time zero to the last sampling time when the concentration was no less than the lower limit of quantification (LLQ). AUC0-t was calculated according to the mixed log-linear trapezoidal rule.
ORR by investigators/IRC per system | Approximately 1 year
  ORR defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Disease Control Rate (DCR) by investigators/IRC per system | Approximately 1 year
  DCR defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) or a stable disease (SD) of 8 weeks or longer based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Duration of Response (DoR) by investigators/IRC per system | Approximately 1 year
  DoR is defined as the time from the date of first documented CR or PR, assessed by investigator and based on RECIST v. 1.1, to the documented date of progressive disease (PD) or death, whichever occurred first.
Progression Free Survival (PFS) by investigators/IRC per system | Approximately 2 years
  PFS defined as the time from the date the participant started study drug to the date the participant experiences an event of disease progression or death.
Overall Survival (OS) | Approximately 2 years
  OS defined as the time from the date the participant started study drug to death for any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Kan Gong, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China